CLINICAL TRIAL: NCT07259564
Title: Phase II Clinical Study of Single Oral Administration of GS3-007a for Oral Suspension in the Diagnosis of AGHD: A Multicenter, Randomized, Open-Label, Three-Way Crossover Trial
Brief Title: A Study of GS3-007a for Oral Suspension in the Diagnosis of Adult Growth Hormone Deficiency (AGHD)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GenSci073-202
Record Dates: First submitted 2025-11-13; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-10

CONDITIONS: Adult Growth Hormone Deficiency (AGHD)
Keywords: adult growth hormone deficiency; GS3-007a dry suspension
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GHST Sequence 1 (Experimental): GS3-007a low dose, GS3-007a high dose, Insulin Tolerance Test
  Interventions: Drug: GS3-007a dry suspension; Drug: Insulin
- GHST Sequence 2 (Experimental): GS3-007a high dose, Insulin Tolerance Test, GS3-007a low dose
  Interventions: Drug: GS3-007a dry suspension; Drug: Insulin
- GHST Sequence 3 (Experimental): Insulin Tolerance Test, GS3-007a low dose, GS3-007a high dose
  Interventions: Drug: GS3-007a dry suspension; Drug: Insulin

INTERVENTIONS:
Drug: GS3-007a dry suspension — GS3-007a dry suspension, low dose body weight, drinking solution, single dose GS3-007a dry suspension, high dose body weight, drinking solution, single dose
  Other Names: GS3-007a
Drug: Insulin — Insulin, 0.10 -0.15 U/kg, intravenous injection, single dose
  Other Names: Insulin Tolerance Test (ITT)

SUMMARY:
The GS3-007a Growth Hormone Stimulation Test (GHST) will be compared with the Insulin Tolerance Test (ITT) in an open-label, randomized, three-way crossover trial. The trial will include subjects suspected to have adult growth hormone deficiency (AGHD) and a group of healthy control subjects.

DETAILED DESCRIPTION:
Trial subjects will be assigned to groups of descending likelihood of having AGHD:

Group A: High likelihood of AGHD Group B: Intermediate likelihood of AGHD Group C: Low likelihood of AGHD Group D: Healthy control subjects matched to Group A. The sequential of the GHSTs for Group A-C will be determined by randomization. Group D will undergo testing in the same sequence as their matched Group A counterparts Serum growth hormone (GH) concentrations will be measured at predefined time points before and after GHST with GS3-007a or insulin. The peak GH value and diagnostic cut-off for GS3-007a dry suspension will be evaluated using receiver operating characteristic (ROC) curves. Safety, pharmacokinetics (PK), and pharmacodynamics (PD) outcomes were assessed for GS3-007a. The Insulin Tolerance Test (ITT) served as the comparator to determine positive and negative agreement with GS3-007a GHSTs.

ELIGIBILITY:
Inclusion Criteria:

Suspected AGHD Subjects (Groups A, B, and C):

* Age ≥ 18 years and ≤ 65 years, male or female.
* Suspected AGHD, meeting at least one of the following criteria:

  * Congenital structural/gene defects in the hypothalamus or pituitary gland, or
  * History of surgery or radiotherapy in the hypothalamic or pituitary region, or
  * Adult traumatic brain injury (TBI) or central nervous system (CNS) infection, or
  * Confirmed deficiency of at least one pituitary hormone other than growth hormone (GH), or
  * Idiopathic childhood-onset GHD.
* IGF-1 SDS < 0.
* Willing and able to comply with the study procedures and voluntarily sign the informed consent form.

Matched Healthy Control Subjects (Group D):

* Age ≥ 18 years and ≤ 65 years, male or female.
* Matching criteria with Group A (subjects with highly suspected AGHD):

  1. Sex;
  2. Age;
  3. BMI;
  4. (If feasible) Estrogen use and administration route (oral, transdermal) in females:

Exclusion Criteria:

* Known or suspected hypersensitivity to growth hormone secretagogues (GHS) or their excipients or known allergy to insulin or its excipients.
* Clinically significant conditions newly diagnosed within 6 months before screening, making the subject unsuitable for ITT:

  1. Chronic congestive heart failure (New York Heart Association (NYHA) Class III or higher);
  2. Other significant cardiovascular/cerebrovascular diseases, e.g., uncontrolled severe hypertension, severe arrhythmia, stroke or transient ischemic attack (TIA), or confirmed coronary artery disease;
  3. Traumatic brain injury (TBI).
* Short-acting GH therapy within 30 days before screening.
* Long-acting GH therapy within 90 days before screening.
* GH stimulation test performed within 7 days before the first dose.
* Abnormal thyroid function during screening, or any adjustment to thyroid hormone replacement therapy dosage prior to the first study dose.
* Abnormal gonadal function during screening, or any adjustment to testosterone/estrogen replacement therapy dosage prior to the first study dose.
* Abnormal adrenal function during screening, or any adjustment to glucocorticoid replacement therapy dosage prior to the first study dose.
* Type 1 diabetes diagnosed before screening, or uncontrolled Type 2 diabetes
* Body mass index (BMI) ≥40.0 kg/m².
* Major surgery (e.g., coronary bypass, hepatectomy/nephrectomy, gynecologic surgery) within 6 months before screening.
* Acute neurological, digestive, respiratory, circulatory, endocrine, or hematologic diseases within 3 months before screening, judged by the investigator to potentially affect drug absorption, distribution, metabolism, excretion (ADME), or safety evaluation.
* History or current diagnosis of malignancy (any type) before screening.
* Electrocardiogram (ECG) findings during screening indicating QTc interval >450 ms, or history of corrected QT interval (QTc) prolongation, or other clinically significant ECG abnormalities, or use of medications known to prolong QTc interval.
* Sellar region MRI scan during screening showing untreated intracranial tumor growth.
* History of clinically symptomatic psychiatric disorders persisting at screening.
* History of Parkinson's disease or epilepsy persisting at screening.
* Females with positive blood human chorionic gonadotropin (hCG) during screening, or lactating females, or females planning pregnancy from screening through follow-up completion.
* Liver function abnormalities during screening
* Use of medications directly affecting pituitary GH secretion or somatostatin-releasing drugs within a period >5 half-lives before first study dose.
* Use of strong cytochrome P450 family 3 subfamily A member 4/5 (CYP3A4/5) inhibitors or inducers.
* Participation in any other drug or medical device clinical trial within 1 month prior to screening, or screening occurring within 5 half-lives of the investigational drug (whichever is longer).
* Unwillingness to use protocol-specified contraception methods
* Other conditions deemed by the investigator to make the subject unsuitable for participation in this clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-19 (Estimated); Primary Completion 2026-05-12 (Estimated); Study Completion 2026-06-09 (Estimated)

PRIMARY OUTCOMES:
ROC curves and the area under the curve (AUC) of the ROC curves | up to 120minutes

SECONDARY OUTCOMES:
Youden index of the ROC curve for GS3-007a dry suspension | up to 120minutes
Number of Participants With Treatment Emergent Adverse Events (TEAEs) | Up to 22 days

OTHER OUTCOMES:
Concentrations of GS3-007a and its metabolite GS3-017 in suspected AGHD subjects | up to 120minutes
Serum GH concentration in suspected AGHD subjects | up to 120minutes
Positive agreement rate, negative agreement rate, and overall agreement rate between GS3-007a dry suspension and ITT in diagnosing AGHD | up to 120minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China